CLINICAL TRIAL: NCT06432335
Title: E-Socket, Diagnostic Monitoring
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Joan E Sanders, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00016676
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Trans-Tibial Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- E-Socket Monitoring (Other)
  Interventions: Other: E-Socket Monitoring

INTERVENTIONS:
Other: E-Socket Monitoring — Limb-socket motion data is collected during participant take-home use. Bimonthly telephone interviews are conducted to assess participant residual limb health status. Analysis is conducted to determine if limb motions and activity changes precede limb health changes.

SUMMARY:
The long-term goal of this research is a socket-embedded prosthesis use and socket fit monitor (E-Socket) that facilitates clinical decision-making in the diagnosis and prognosis of health issues faced by people with transtibial amputation. The overall strategy is to enhance the E-socket to include additional metrics that we identified needed from studies to date (Aim #1). Then we conduct a randomized control trial testing the diagnostic utility of the E-socket data in clinical care (Aim #2). From the data collected in that study, we develop the prognostic capability of the system (Aim #3).

Aim 3 will not involve human subject testing as it will focus on the development of the system in preparation for a future aim involving participants' own clinicians.

Note: we use the term "diagnostic" throughout our application in a general sense. The device will not be diagnosing specific diseases or medical conditions.

ELIGIBILITY:
Inclusion Criteria:

-

Prosthesis Users:

Aims 1 and 2

* Over 18 years of age
* Unilateral or bilateral trans-tibial amputation at least 12 months prior
* Have a limb of length 9 cm or greater
* Are capable of at least 5 minutes of continuous walking
* Regularly use a definitive prosthesis
* Do not regularly use assistive devices (e.g., cane, walker) for ambulation
* Do not have open wounds on their residual limb at the time of enrollment

Aim 2

-Regularly visit their prosthetist at least twice a year,

Exclusion Criteria:

-

Prosthesis Users:

Aims 1 and 2

* Reduced skin sensation
* Presence of skin breakdown
* Regular use of an assistive device
* Persons with trans-femoral amputation

Aim 1 Only

-Vacuum suspension users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Anterior-Distal Limb Motion | 12 months
  Monitor anterior-distal limb motion in the prosthesis to determine if limb motions and activity changes precede changes in limb health. Interviews with the participants and questionnaires will be used to assess the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sanders, Principal Investigator — University of Washington